

# STATISTICAL ANALYSIS PLAN

### ALK22/ENZ215-DEN1

A randomized, double-blind, three-arm, parallel-group, single-dose study to compare the pharmacokinetics, pharmacodynamics, safety, tolerability, and immunogenicity of Denosumab (ENZ215, EU-sourced Prolia®, and US-sourced Prolia®) in healthy adult male volunteers

**AUTHOR:** ASHUTOSH RANJAN, PIYUSHKUMAR JOGANI

**VERSION NUMBER AND DATE:** V1.0, 21JUN2024

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP

Author: Ashutosh Ranjan, Piyushkumar Jogani Version Number: 1.0

Version Date: 21JUN2024

Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V1.0 (Dated 21JUN2024) for Protocol ALK22/ENZ215-DEN1.

| | Name | Signature | Date (DDMmmYYYYY) |
|---|---|---|---|
| Author: | Ashutosh Ranjan | DocuSigned by Ashutosh Ra | June 24, 2024<br>anjan |
| Position: | Statistical Scientist | A SILLIFACIL P. A. A | am the author of this document<br>une 24, 2024 2:35:50 PM BST |
| Company: | IQVIA | 55DBAAC88C76431C85522 | 29B736B6AF8D |
| Author: | Piyushkumar Jogani | DocuSigned by Piyushkuma | i Jogani June 24, 2024 |
| Position: | Biostatistician, Biostati | 1 Prigustalammang Jogan | June 24, 2024 5:22:53 AM EDT |
| Company: | Premier Research | D1E3500D6D854D0380A0I | B51EE2459E48 |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (D | DMmmYYYY) |
|---|---|---|---|---|
| Approved By: | Dr. Vinayaka Shahavi | DocuSigned by Vinayak | a Shahavi | June 22, 2024 |
| Position: | General Manager – Clinic | s <b>viinl</b> ayaka Sha | ahavi | I approve this document<br>June 22, 2024 12:03:55 |
| Company: | Alkem Laboratories Ltd. | D3E46A69468042D8B9 | 8B6A970A59 | 9FD0A |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Statistical Analysis Plan 

## **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 21JUN2024) for Protocol ALK22/ENZ215-DEN1.

| | Name | | Signature | Date (DDMmmYYYY | | <b>(</b> ) | |
|---|---|---|---|---|---|---|---|
| Author: | Ashutosh Ranjan | | DocuSigned by Ashutos | | ne 2 | | 202 |
| Position: | Statistical Scientist | V | Ashvtosh Panjan | î the author of this doo<br>e 24, 2024 2:36:07 F | | | |
| Company: | IQVIA | | -55DBAAC88C76431C855229B736B6AF8D | | | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMmmYYYY) |
|---|---|---|---|
| Approved By: | Dr. Vinayaka Shahavi | DocuSigned by Vinayaka | |
| Position: | General Manager – Clinic | s <b>Vana</b> yaka Sha | havi lapprove this document June 22, 2024 12:04:58 AM PD7 |
| Company: | Alkem Laboratories Ltd. | D3E46A69468042D8B9 | 8B6A970A59FD0A |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


## **MODIFICATION HISTORY**

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| 1.0 | 21JUN2024 | Ashutosh Ranjan, | Not Applicable – First Version |
| | | Piyushkumar Jogani | |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



## **TABLE OF CONTENTS**

| l. | INTRODUCTION | 11 |
|------|-------------------------------------|----|
| 2. | STUDY OBJECTIVES | 11 |
| 2.1. | Primary Objective | 11 |
| 2.2. | Secondary Objectives | 11 |
| 3. | STUDY ENDPOINTS | 11 |
| 3.1. | Primary Endpoints | 11 |
| 3.2. | Secondary Endpoints | 17 |
| 3.2 | v i | |
| 3.2 | | |
| 3.2 | 2.3. Safety | 12 |
| 4. | STUDY DESIGN | 12 |
| 4.1. | General Description | 12 |
| 4.2. | Schedule of Events | 14 |
| 4.3. | Changes to Analysis from Protocol | 14 |
| 5. | PLANNED ANALYSES | 14 |
| 5.1. | Final Analysis | 14 |
| 6. | ANALYSIS SETS | 14 |
| 6.1. | Process for Analysis Set Assignment | 14 |
| 6.2. | All Subjects Randomized Set [RAN] | 15 |
| 6.3. | Safety Analysis Set [SAF] | 15 |
| 6.4. | Pharmacokinetic Analysis Set [PKAS] | 15 |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



| Sta | Statistical Analysis Plan | |
|-------|--------------------------------------------------------|----|
| 6.5. | Pharmacodynamic Analysis Set [PDAS] | 15 |
| 7. | GENERAL CONSIDERATIONS | 15 |
| 7.1. | Summary Statistics | 15 |
| 7.2. | Treatment Summarization | 16 |
| 7.3. | Precision | 16 |
| 7.4. | Reference Start Date and Study Day | 17 |
| 7.5. | Baseline | 19 |
| 7.6. | Retests, Unscheduled Visits and Early Termination Data | 19 |
| 7.7. | Statistical Tests | 19 |
| 7.8. | Common Calculations | 20 |
| 7.9. | Software Version | 20 |
| 8. | STATISTICAL CONSIDERATIONS | 20 |
| 8.1. | Missing Data | 20 |
| 9. | OUTPUT PRESENTATIONS | 21 |
| 10. | DISPOSITION AND WITHDRAWALS | 21 |
| 11. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 21 |
| 12. | PROTOCOL DEVIATIONS | 22 |
| 12.1. | Deviations Related to Study Conduct | 22 |
| 12.2. | Deviations Related to PK and PD Analysis | 22 |
| 13. | SURGICAL AND MEDICAL HISTORY | 22 |
| 14. | MEDICATIONS | 22 |

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-Document:

DEN1\_HAB89093\Biostatistics\Documentation\SAP

1.0 Author: Ashutosh Ranjan, Piyushkumar Jogani Version Number:

STUDY MEDICATION EXPOSURE ......23

PHARMACOKINETIC ANALYSIS......23


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

**15.** 

**16.** 



| Statistical | Analy | vsis | Plan |
|-------------|-------|------|------|
|-------------|-------|------|------|

| 16.2. Pharmacokinetic Parameters | 16.1. | Serum Concentration Data | | 23 |
|---|---|---|---|---|
| 17.1. Pharmacodynamic Concentrations 17.2. Pharmacodynamic Parameters | 16.2. | Pharmacokinetic Parameters | | 24 |
| 17.2. Pharmacodynamic Parameters | 17. P | HARMACODYNAMIC ANALYSIS | | 27 |
| 18. SAFETY OUTCOMES | 17.1. | Pharmacodynamic Concentrations | | 27 |
| 18.1. Adverse Events | 17.2. | Pharmacodynamic Parameters | | 28 |
| 18.1.1. All TEAEs 18.1.1.1. Severity 18.1.1.2. Relationship to Study Medication 18.1.3. Serious Adverse Events 18.1.4. Injection Site Reaction Assessment 18.2. Deaths 18.3. Laboratory Evaluations 18.3.1. Laboratory Reference Ranges 18.4. ECG Evaluations 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS 1QVIA Output Conventions Document: \\dccar2dnetynasc01p-lan1.quintiles.net\cp_ops\BlOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | 18. S. | AFETY OUTCOMES | | 29 |
| 18.1.1.1 Severity. 18.1.1.2 Relationship to Study Medication. 18.1.2. TEAES Leading to Discontinuation of Study Medication. 18.1.3. Serious Adverse Events. 18.1.4 Injection Site Reaction Assessment. 18.2 Deaths. 18.3 Laboratory Evaluations. 18.3.1 Laboratory Reference Ranges. 18.4. ECG Evaluations. 18.4.1 Clinically Noteworthy ECG Criteria. 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES | | | | |
| 18.1.1.2. Relationship to Study Medication 18.1.2. TEAEs Leading to Discontinuation of Study Medication 18.1.3. Serious Adverse Events 18.1.4. Injection Site Reaction Assessment 18.2. Deaths 18.3. Laboratory Evaluations 18.3.1. Laboratory Reference Ranges 18.4. ECG Evaluations 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS 1QVIA Output Conventions Document: \\dccar2dnetynasc01p-lan1.quintiles.net\cdot\cdotcp-ops\BIOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | - | | | |
| 18.1.2 TEAEs Leading to Discontinuation of Study Medication 18.1.3. Serious Adverse Events 18.1.4. Injection Site Reaction Assessment 18.2. Deaths 18.3. Laboratory Evaluations 18.3.1. Laboratory Reference Ranges 18.4. ECG Evaluations 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 18.9. Immunogenecity Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS IQVIA Output Conventions. Document: \\dccar2dnetynasc01p-lan1.quintiles.net\cdot\cdot\cdot\cdot\cdot\cdot\cdot\cdo | | 3 | | |
| 18.1.3. Serious Adverse Events 18.1.4. Injection Site Reaction Assessment 18.2. Deaths 18.3. Laboratory Evaluations 18.3.1. Laboratory Reference Ranges 18.4. ECG Evaluations 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 18.9. Immunogenecity Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS IQVIA Output Conventions. Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cdotcp_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | | | | |
| 18.1.4. Injection Site Reaction Assessment 18.2. Deaths 18.3. Laboratory Evaluations 18.3.1. Laboratory Reference Ranges 18.4. ECG Evaluations 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 18.9. Immunogenecity Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS IQVIA Output Conventions Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | | | | |
| 18.2. Deaths 18.3. Laboratory Evaluations 18.3.1. Laboratory Reference Ranges 18.4. ECG Evaluations 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs 18.6. Physical Examination 18.7. Oral Examination 18.8. COVID-19 Assessment 18.9. Immunogenecity Assessment 19. DATA NOT SUMMARIZED OR PRESENTED 20. REFERENCES APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS IQVIA Output Conventions Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cdot\cdot\cdot\cdot\cdot\cdot\cdot\cdo | | | | |
| 18.3.1. Laboratory Reference Ranges | 18.2. | · | | |
| 18.3.1. Laboratory Reference Ranges | 18.3. | Laboratory Evaluations | | 3 |
| 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs | | | | |
| 18.4.1. Clinically Noteworthy ECG Criteria 18.5. Vital Signs | 10.4 | ECC E al. d'ann | | 2/ |
| 18.5. Vital Signs | | | | |
| 18.6. Physical Examination | 10.4.1. | Chilically Noteworthy ECG Criteria | | |
| 18.7. Oral Examination | 18.5. | Vital Signs | | 33 |
| 18.7. Oral Examination | 18 6 | Physical Examination | | 33 |
| 18.8. COVID-19 Assessment | 10.0. | 1 Hysical Examination | | |
| 18.9. Immunogenecity Assessment | 18.7. | Oral Examination | | 33 |
| 18.9. Immunogenecity Assessment | 10.0 | COLUMN 40. | | |
| 19. DATA NOT SUMMARIZED OR PRESENTED | 18.8. | COVID-19 Assessment | •••••• | 33 |
| 20. REFERENCES | 18.9. | Immunogenecity Assessment | | 34 |
| 20. REFERENCES | | | | |
| 20. REFERENCES | 19. D | ATA NOT SUMMARIZED OR PRESENT | ΓΕD | 32 |
| APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | | | | |
| IQVIA Output Conventions Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | | | | |
| Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | APPEN | DIX 1. PROGRAMMING CONVENTION | ONS FOR OUTPUTS | |
| Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-DEN1_HAB89093\Biostatistics\Documentation\SAP | IQVIA C | Output Conventions | | 30 |
| _ | | t: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\\ | BIOS\Alkem\Denosumab\ALK22EN | |
| Addition Administry Type There are a few and the American Techniques and the American | Author: | <del>-</del> | | 1.0 |
| Version Date: 21JUN2024 | | | | 21JUN2024 |

Effective Date: 01Nov2021

Template No.: CS\_TP\_BS016 Revision 7

Reference: CS\_WI\_BS005



| Page | 8 | of | 4 | 1 |
|------|---|----|---|---|
|------|---|----|---|---|

| Dates & Times | 36 |
|------------------------------------------------------|--------------|
| Spelling Format | 36 |
| Presentation of Treatment Groups | 36 |
| Presentation of Visits | 36 |
| Listings | 36 |
| APPENDIX 2. PARTIAL DATE CONVENTIONS | 37 |
| Algorithm for Treatment Emergence of Adverse Events: | 37 |
| Algorithm for Prior / Concomitant Medications: | 38 |
| APPENDIX 3. SAFETY LABORATORY CONVERSION FACTOR | AND UNITS 40 |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




## LIST OF ABBREVIATIONS

| ABBREVIATION | TERM |
|---|---|
| ADAs | Antidrug antibodies |
| AE | Adverse Event |
| ANCOVA | Analysis of covariance |
| AUC <sub>0-inf</sub> | Area under the drug concentration-time curve from time 0 to infinity |
| AUC <sub>0-t</sub> | Area under the drug concentration-time curve from day 0 to day 270 |
| AUC <sub>0 - Day 28</sub> | Partial area under the drug concentration-time curve from time 0 (pre-dose) to day 28 |
| AUEC | Area under the effect curve from time 0 to day 270 |
| BMI | Body mass index |
| C <sub>max</sub> | Maximum observed drug concentration |
| CI | Confidence Interval |
| CL/F | Apparent systemic clearance |
| COVID-19 | Coronavirus disease 2019 |
| CTX-1 | C-terminal telopeptide type-1 |
| CV | Coefficient of variation |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EOS | End of Study |

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-Document:

DEN1\_HAB89093\Biostatistics\Documentation\SAP

1.0 Author: Ashutosh Ranjan, Piyushkumar Jogani Version Number:


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

 $Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 \ IQVIA. \ All \ rights \ reserved. \ The \ contents \ of this \ document \ are \ confidential \ and \ proprietary \ to \ IQVIA \ Holdings \ Inc. \ and \ its \ subsidiaries. \ Unauthorized \ use, \ disclosure \ or \ reproduction \ is \ strictly \ prohibited.$ 




| EU | European Union |
|------------------|-------------------------------------------------|
| mL | Milliliter |
| NAB | Neutralizing antibodies |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| SAE | Serious Adverse Event |
| SARS-CoV- 2 | Severe acute respiratory syndrome coronavirus-2 |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| T <sub>max</sub> | Time to reach C <sub>max</sub> |
| $T_{1/2}$ | Terminal elimination half-life |
| ULN | Upper Limit of Normal |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



#### 1. Introduction

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of safety, pharmacokinetic (PK), pharmacodynamic (PD), and immunogenicity data for Protocol ALK22/ENZ215-DEN1. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This SAP is based on protocol version 4.0, dated 03OCT2022.

### 2. STUDY OBJECTIVES

## 2.1. Primary Objective

The primary objective is to demonstrate bioequivalence between ENZ215 and EU- and US-sourced Prolia® using PK parameters.

## 2.2. Secondary Objectives

The secondary objectives are:

To compare the serum PK profile of ENZ215 and EU- and US-sourced Prolia®

- To compare the serum CTX-1 profile of ENZ215 and EU- and US-sourced Prolia®
- To compare the immunogenicity profile of ENZ215 and EU- and US-sourced Prolia®
- To compare the safety and tolerability profile of ENZ215 and EU- and US-sourced Prolia®

#### 3. STUDY ENDPOINTS

# 3.1. Primary Endpoints

The primary endpoints are maximum observed drug concentration ( $C_{max}$ ), area under the drug concentration-time curve from day 0 to day 270 (AUC<sub>0-t</sub>) and area under the drug concentration-time curve from time 0 to infinity (AUC<sub>0-inf</sub>) of ENZ215 and EU- and US-sourced Prolia®.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


# 3.2. Secondary Endpoints

#### 3.2.1. Pharmacokinetics

The secondary PK endpoints are:

- Partial area under the drug concentration-time curve from time 0 (pre-dose) to day 28
- Time to reach C<sub>max</sub> (t<sub>max</sub>)
- Terminal elimination half-life  $(t_{1/2})$
- Apparent systemic clearance (CL/F)

## 3.2.2. Pharmacodynamics

The secondary PD endpoint is area under the effect curve (AUEC) from time 0 to Day 270 for serum CTX-1 percent inhibition:

### **3.2.3.** Safety

The secondary safety endpoints are:

- Number of subjects who developed denosumab neutralizing antibodies and antidrug antibodies (Day 1, 28, 90, 180, and 270)
- Incidence of adverse events
- Clinically significant changes in physical examination findings, safety laboratory analyses (serum chemistry, hematology, and urinalysis), vital signs, and 12-lead electrocardiogram (ECG)

### 4. STUDY DESIGN

# 4.1. General Description

This is a randomized, double-blind, three-arm, parallel-group, single-dose study to demonstrate bioequivalence of ENZ215 and EU- and US-sourced Prolia after a single 60-mg dose administered subcutaneously in healthy adult male volunteers.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




Subjects will be screened for enrolment in the study from day -28 to day -1 before randomization. Approximately 207 subjects will be enrolled into 3 groups (69 in each group) in parallel. The subjects may be enrolled in multiple groups at the site. All the eligible subjects will be randomized (1:1:1) to receive a single SC 60-mg dose of either ENZ215 or EU- or US-sourced Prolia on Day 0/1.

Eligible subjects will be admitted/check-in to the phase 1 study site at least 10 hours prior to dosing on day 1 and will be discharged/check out from phase 1 study site on day 2 after PK sample collection (in-subject period).

All screening and on-study blood samples will be processed and sent to local or central laboratory as applicable as defined in the lab manual. Further details on study design are provided in Section 8.1 of study protocol.

Table 1 Study Flow Chart



End of Study (EoS) assessment will be performed on Day 270 (week 39) or at the time of early discontinuation/withdrawal of the subject.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Statistical Analysis Plan 

#### 4.2. Schedule of Events

Schedule of events can be found in Section 5.2 of the protocol.

## 4.3. Changes to Analysis from Protocol

Not applicable.

#### 5. PLANNED ANALYSES

Final analysis following database lock will be performed for this study.

## 5.1. Final Analysis

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics and Premier Research Group (India) Private Limited following Sponsor Authorization of this Statistical Analysis Plan, identification of major protocol deviations requiring analysis exclusions, Database Lock, determination of analysis sets and Unblinding of Treatment.

#### 6. ANALYSIS SETS

Agreement and authorization of subjects included/excluded from each analysis set will be conducted prior to the unblinding of the study.

# 6.1. Process for Analysis Set Assignment

Agreement and authorization regarding participants included/excluded from the PK/PD analysis population will be achieved prior to the final database hard lock, once the Premier Research team creates the list of subjects that need to be excluded from the PK/PD population. Before the database lock, the sponsor will review the list of all participants to be excluded from the pertinent analysis populations, along with the reasons for their exclusion from the analysis populations and provide approval/confirmation.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




#### 6.2. All Subjects Randomized Set [RAN]

The all subjects randomized (RAN) set will contain all subjects who were randomized to study treatment.

#### 6.3. Safety Analysis Set [SAF]

The safety analysis set (SAF) will contain all subjects who received the single dose of the study drug and subjects will be classified according to treatment received.

#### 6.4. Pharmacokinetic Analysis Set [PKAS]

All subjects who comply sufficiently with the protocol who received the single dose of the study drug and had one pre-dose and at least one post-dose measurement of any of the PK assessment not impacted by any protocol deviations.

#### 6.5. Pharmacodynamic Analysis Set [PDAS]

All subjects who comply sufficiently with the protocol, who received the single dose of the study drug and had one pre-dose and at least one post-dose measurement of any of the PD assessment.

### 7. GENERAL CONSIDERATIONS

Derivation of the PK and PD parameters for Denosumab in serum will be the responsibility of the clinical pharmacokineticist at Premier Research Group (India) Private Limited. The PK, PD and Immunogenicity summaries (tables and figures) and data listings as well as the datasets including ADaM for PK, PD and Immunogenicity will be the responsibility of the study biostatistician at Premier Research Group (India) Private Limited, whereas the SDTM dataset for PC/PP and IS will be developed by IQVIA. The safety summaries (tables) and data listings will be the responsibility of the study biostatistician at IQVIA.

#### 7.1. **Summary Statistics**

For qualitative variables, the population size (N for sample size and n for available data) and the percentage (of available data) for each class of the variable will be presented. Quantitative variables will

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-Document:

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Reference: CS\_WI\_BS005 Template No.: CS\_TP\_BS016 Revision 7

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

be summarized using descriptive statistics, including N, n, mean, standard deviation (SD), coefficient of variation (CV%), median, minimum, and maximum values. Coefficient of variation will not be presented for change from baseline results.

Pharmacokinetic concentrations and parameters will be summarized using N, n, mean, SD, coefficient of variation (CV%), median, minimum and maximum. Statistics for PK parameters [except for time to reach  $C_{max}$  ( $t_{max}$ )] will additionally include geometric mean (GM) and geometric CV% (GCV%). The  $t_{max}$  will be summarized with N, n, median, minimum, and maximum only.

Pharmacodynamic serum CTX-1 estimation and parameters will be summarized using N, n, mean, SD, coefficient of variation (CV%), median, minimum and maximum. Statistics for PD parameters will additionally include geometric mean (GM) and geometric CV% (GCV%).

Further details of summarization of PK and PD variables are discussed in Section 16 and 17.

#### 7.2. Treatment Summarization

In general, data will be presented by treatment. Data for all study subjects combined will also be presented when appropriate.

#### 7.3. Precision

Safety variables (i.e., clinical laboratory values, vital signs, and ECG intervals), including derivations thereof, will be reported to the same precision as the source data.

All PK concentrations and pharmacodynamic results will be reported and analyzed to 3 significant digits. Derived PK and PD parameters will be rounded for reporting purposes in by-subject listings. The unrounded derived PK and PD data will be considered the source data for the calculation of descriptive statistics and the statistical analysis. For most derived PK (i.e. AUC<sub>0-t</sub>, AUC<sub>0-inf</sub>, AUC<sub>0-Day 28</sub>, T<sub>1/2</sub>, CL/F) and PD parameters (i.e. AUEC), 3 significant digits will be used as the standard rounding procedure, with the following exceptions:

• Parameters directly derived from source data (i.e., C<sub>max</sub> will be reported and analyzed with the same precision as the source data.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




• Parameters derived from actual elapsed sample collection times (eg, t<sub>max</sub>) will be reported with the same precision as the actual elapsed sampling time value of the source data.

For the reporting of descriptive statistics, the mean, SD, standard error and confidence intervals (CIs) will be presented to one digit more precision than the source data. The minimum, median, and maximum will be presented to the same precision as the source data. Coefficient of variation and GeoCV% will always be reported to 1 decimal place. Ratios of means for PK and PD parameters and their associated CIs will be presented with two decimal places (as a percentage) to meet regulatory requirements. A minimum of n=3 is required for all descriptive statistics to be generated. If n is less than 3, only N, n, minimum and/or maximum will be reported, as appropriate. P-values, if any, shall be reported to four decimal places or as <0.0001.

## 7.4. Reference Start Date and Study Day

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and events.

Reference start date is defined as the day of the first study medication administration (Day 1) and Study Day will be determined as:

- If the date of the event is on or after the reference date, then: Study Day = (date of event reference date) + 1.
- If the date of the event is prior to the reference date, then: Study Day = (date of event reference date).

In the situation where the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the listings.

The PK sample window rule is as follows:

| Nominal study Time point | Window<br>Period | Lower Upper | | Target<br>Time (h) |
|---|---|---|---|---|
| 0 hour (pre-dose) | NA | NA | NA | NA |
| Day 1 (1 hours) | ± 10 minutes | 50 minutes | 70 minutes | 1 |
| Day 1 (4 hours) | ± 10 minutes | 230 minutes | 250 minutes | 4 |
| Day 1 (8 hours) | ± 10 minutes | 470 minutes | 490 minutes | 8 |
| Day 1 (12 hours) | ± 10 minutes | 710 minutes | 730 minutes | 12 |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


| Nominal study Time point | Window<br>Period | Lower | Upper | Target<br>Time (h) |
|---|---|---|---|---|
| Day 2 (24 hours) | ± 10 minutes | 1450 minutes | 1430 minutes | 24 |
| Day 3 (48 hours) | ± 2 hours | 46 hours | 48 hours | 48 |
| Day 4 (72 hours) | ± 2 hours | 70 hours | 74 hours | 72 |
| Day 5 (96 hours) | ± 2 hours | 94 hours | 98 hours | 96 |
| Day 6 (120 hours) | ± 2 hours | 118 hours | 122 hours | 120 |
| Day 8 (168 hours) | ± 2 hours | 166 hours | 170 hours | 168 |
| Day 10 (216 hours) | ± 2 hours | 214 hours | 218 hours | 216 |
| Day 12 (264 hours) | ± 2 hours | 262 hours | 266 hours | 264 |
| Day 16 (360 hours) | ± 2 hours | 358 hours | 362 hours | 360 |
| Day 21 (480 hours) | ± 2 hours | 478 hours | 482 hours | 480 |
| Day 28 (648 hours) (week 4) | ±1 day | 27 days | 29 days | 648 |
| Day 42 (984 hours) (week 6) | ±3 days | 39 days | 45 days | 984 |
| Day 63 (1488 hours) (week 9) | ±3 days | 60 days | 66 days | 1488 |
| Day 90 (2136 hours) (week 13) | ±3 days | 87 days | 93 days | 2136 |
| Day 119 (2832 hours) (week 17) | ±3 days | 116 days | 122 days | 2832 |
| Day 147 (3504 hours) (week 21) | ±3 days | 144 days | 150 days | 3504 |
| Day 180 (4296 hours) (week 26) | ±3 days | 177 days | 183 days | 4296 |
| Day 224 (5352 hours) (week 32) | ±5 days | 219 days | 229 days | 5332 |
| Day 270 (6456 hours) (week 39) (EOS) | ±5 days | 265 days | 275 days | 6456 |

If any sample will be collected out of window period it will be considered as deviation and actual sample collection time will be used in the PK analysis.

The PD sample window rule is as follows:

| Nominal study Time point | Window<br>Period | Lower | Upper | Target<br>Time (h) |
|---|---|---|---|---|
| 0 hour (pre-dose) | NA | NA | NA | NA |
| Day 2 (24 hours) | ± 10 minutes | 1450 minutes | 1430 minutes | 24 |
| Day 3 (48 hours) | ± 2 hours | 46 hours | 48 hours | 48 |
| Day 4 (72 hours) | ± 2 hours | 70 hours | 74 hours | 72 |
| Day 5 (96 hours) | ± 2 hours | 94 hours | 98 hours | 96 |
| Day 6 (120 hours) | ± 2 hours | 118 hours | 122 hours | 120 |
| Day 8 (168 hours) | ± 2 hours | 166 hours | 170 hours | 168 |
| Day 10 (216 hours) | ± 2 hours | 214 hours | 218 hours | 216 |
| Day 12 (264 hours) | ± 2 hours | 262 hours | 266 hours | 264 |
| Day 16 (360 hours) | ± 2 hours | 358 hours | 362 hours | 360 |
| Day 21 (480 hours) | ± 2 hours | 478 hours | 482 hours | 480 |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


| Nominal study Time point | Window<br>Period | Lower | Upper | Target<br>Time (h) |
|---|---|---|---|---|
| Day 28 (648 hours) (week 4) | ±1 days | 27 days | 29 days | 648 |
| Day 63 (1488 hours) (week 9) | ±3 days | 60 days | 66 days | 1488 |
| Day 119 (2832 hours) (week 17) | ±3 days | 116 days | 122 days | 2832 |
| Day 180 (4296 hours) (week 26) | ±3 days | 177 days | 183 days | 4296 |
| Day 270 (6456 hours) (week 39) (EOS) | ±5 days | 265 days | 275 days | 6456 |

If any sample will be collected out of window period it will be considered as deviation and actual sample collection time will be used in the PD analysis.

#### 7.5. Baseline

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments) and will correspond to Screening value for ECG and safety laboratory assessments, and to Day 1 predose for vital signs, PD and albumin-adjusted calcium.

### 7.6. Retests, Unscheduled Visits and Early Termination Data

Unscheduled measurements will not be included in summary statistics but will contribute to the assessment of clinical outliers where applicable. Early termination results will be recorded as such and included with the end of study summaries.

In the case of a retest of a scheduled assessment, the earliest available measurement for that scheduled time (i.e., the original assessment) will be used for summaries unless flagged as invalid.

Listings will include all scheduled, unscheduled, retest, and early discontinuation data.

#### 7.7. Statistical Tests

The default significant level will be (5%); confidence intervals will be 90% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


### 7.8. Common Calculations

For quantitative safety measurements, change from baseline will be calculated as:

- Test Value at Visit X Baseline Value
- Change from baseline (CHG) = Post-baseline Value Baseline Value

For PK computations, the CV%, GM and GCV% will be computed as below:

• 
$$CV\% = 100 * \frac{SD}{mean}$$

•  $GM = e^{Mean_{Log}}$ 

• GCV% = 
$$(100) * \sqrt{e^{SD_{Log}^2}} - 1$$

For the qualitative immunogenicity data will be described as n(%) for respective visit.

#### 7.9. Software Version

All analyses will be conducted using SAS version 9.4 or higher. All derivations, statistical analyses, summaries and listings will be generated using SAS version 9.4 or higher (SAS Institute, Inc., Cary, North Carolina). Non-compartmental pharmacokinetic and pharmacodynamic parameter calculations will be performed using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> 8.3 or higher (Certara, Princeton, New Jersey). Graphics may be prepared using the same versions of SAS.

## 8. STATISTICAL CONSIDERATIONS

## 8.1. Missing Data

Missing safety data will not be imputed.

Missing PK and PD data will be handled as described in section 16.2 and 17.2 of this analysis plan. If any sample data will not be transferred from the bio-analytical lab then it will be considered as missing sample for PK and PD analysis.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




### 9. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs. The mock shells provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by Premier Research Group (India) Private Limited and IQVIA Biostatistics.

The PK, PD and immunogenicity mock shells to be provided by Premier Research Group (India) Private Limited.

Some minor modifications may be necessary to the planned design of tables, figures and listings to accommodate data collected during the actual study conduct.

### 10. DISPOSITION AND WITHDRAWALS

All subjects who are randomized will be accounted for in this study. Subject disposition will be tabulated for each study treatment and for all subjects combined with the number of subjects who are dosed, complete the study, prematurely discontinue, and the reason for early discontinuation. A listing will present dates of completion or early withdrawal and the reason for early discontinuation, if applicable, for each subject.

Listings of study eligibility, treatment randomization, and study treatment administration will be provided.

## 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Individual subject demographics and baseline characteristics (medical/surgical history and results from drug and alcohol screens, cotinine test, and serology screening) will be presented in listings.

Demographic characteristics such as age, sex, race, ethnicity, height, weight, and body mass index (BMI) will be summarized and tabulated by treatment and for all subjects overall. Descriptive statistics will be presented for age, height, weight, and BMI. Frequency counts and percentages will be presented for sex, race, and ethnicity. No statistical testing will be carried out for demographic or other baseline

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




characteristics.

#### **12**. PROTOCOL DEVIATIONS

## 12.1. Deviations Related to Study Conduct

A deviation from a protocol occurs when Investigator site staff or a study subject does not adhere to the protocol's stipulated requirements, whether inadvertently or planned. Protocol deviations will be listed and will include a classification of minor or major, as determined by clinical staff.

Protocol deviations will be reviewed by the study pharmacokineticist, sponsor medical monitor, IQVIA medical monitor and biostatistician prior to unblinding to identify deviations which have the potential to affect the pharmacokinetic or pharmacodynamic results.

## 12.2. Deviations Related to PK and PD Analysis

Based on case-by-case review, Changes to the procedures or events, which may impact the quality of the PK and PD data, will be considered important protocol deviations, and will be described within the clinical study report. These changes or events will include any circumstances that will alter the evaluation of the PK and PD. Examples include, but may not be limited to, inaccurate dosing on the day of PK sampling. Other changes to the procedures or events which do not impact the quality of the PK and PD data will not be considered important protocol deviations. A common example of a non-significant protocol deviation is a missed blood sample or deviations from blood collection times.

#### 13. SURGICAL AND MEDICAL HISTORY

Surgical and medical history, coded using Medical Dictionary for Regulatory Activities (MedDRA), the latest version, will be listed for the safety analysis set.

#### 14. **MEDICATIONS**

Medication usage, coded using the World Health Organization (WHO) Drug Dictionary, the latest version, will be categorized as Prior or Concomitant and listed for the safety population:

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-Document:

DEN1\_HAB89093\Biostatistics\Documentation\SAP

Author: Version Number: 1.0 Ashutosh Ranjan, Piyushkumar Jogani


Reference: CS\_WI\_BS005 Template No.: CS TP BS016 Revision 7

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


- 'Prior' medications are medications which started and stopped prior to the administration of study medication.
- 'Concomitant' medications are medications which were taken during the treatment period, or specifically:
  - o started on or after the administration of study medication
  - started prior to the administration of study medication and were continued after the administration of study medication

See Appendix 2 for handling of partial dates for medications. In the case where it is not possible to define a medication as prior or concomitant, the medication will be classified as concomitant.

#### 15. STUDY MEDICATION EXPOSURE

Exposure to study medication will be listed for the safety analysis set.

### 16. PHARMACOKINETIC ANALYSIS

#### 16.1. Serum Concentration Data

Subjects with partial data will be evaluated on a case-by-case basis to determine if sufficient data are available for reliable estimation of PK parameters. A listing of PK blood sample collection times as well as derived sampling time deviations will be provided.

Serum concentrations of denosumab will be summarized using descriptive statistics for each treatment Concentrations that are below the lower limit of quantification (BLQ) will be treated as zero for the computation of descriptive statistics.

Figures of arithmetic mean concentration-time data (±SD, as appropriate) will be presented for each treatment on linear and semi-logarithmic scales. Individual subject concentration-time data will be graphically presented on linear and semi-logarithmic scales for each treatment. Individual concentrations which are BLQ will be displayed as zero in the graphic presentations on linear scale; but will not be plotted on semi-logarithmic scale. Mean values BLQ will be displayed as 0 in the graphic presentations on linear scale but will not be plotted on semi-logarithmic scale.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




#### 16.2. Pharmacokinetic Parameters

For PK parameter calculations, predose samples that are BLQ will be assigned a numerical value of zero. Any anomalous (quantifiable) concentration values observed at predose will be identified in the study report and used for the computation of PK parameters. The parameters resulting from such an anomalous concentration value will be determined on a case-by-case basis as to whether they will be included in descriptive analyses as well as in Primary endpoint analysis.

Actual elapsed time from dosing will be used if a sample is collected outside the time-window period otherwise scheduled time will be used for the final serum PK parameter calculations.

Any other BLQ concentrations will be assigned a value of zero if they precede quantifiable samples in the initial portion of the profile. A BLQ value that occurs between quantifiable data points, especially prior to  $C_{max}$ , will be assigned a concentration of zero. Following  $C_{max}$ , BLQ values embedded between 2 quantifiable data points will be set to missing when calculating PK parameters. If a BLQ value occurs at the end of the collection interval (after the last quantifiable concentration), it will be set to zero.

#### Pharmacokinetic exclusion criteria:

- No value for AUC<sub>0-inf</sub>, CL/F or T<sub>1/2</sub> will be reported for cases that do not exhibit a terminal log-linear phase in the concentration-time profile.
- Criteria for exclusion of pharmacokinetic parameters of a particular subject will be as below:
  - Three consecutive missing (M) / Non-Reportable (NR) samples in elimination phase may significantly influence the AUC<sub>0-t</sub>, AUC<sub>0-Day 28</sub> and elimination phase dependent parameters (AUC<sub>0-inf</sub> and T<sub>1/2</sub>, CL/F). Inclusion of such parameters in the statistical analysis may mislead the final outcome. Hence, AUC<sub>0-t</sub>, AUC<sub>0-Day 28</sub> and elimination phase dependent parameters (AUC<sub>0-inf</sub> and T<sub>1/2</sub>) will be excluded.
  - Additionally, any subject with at least 3 consecutive Missing (M) / Non-reportable (NR) samples during the absorption phase such subject will be excluded from the pharmacokinetic and statistical analysis. In such a scenario, only plasma concentration versus time data of that subject will be tabulated and reported in the study report.
  - Subjects without measurable concentrations or who have only very low serum concentrations from the reference medicinal product will be excluded from the pharmacokinetic and statistical analyses for the assessment of bioequivalence. A

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


- subject is considered to have very low serum concentrations if his/her AUC is less than 5% of reference medicinal product geometric mean AUC, calculated without inclusion of data from the outlying subject.
- AUC<sub>0-t</sub>/AUC<sub>0-inf</sub> is found to be <0.80 with R<sup>2</sup> adjusted < 0.80 for Kel estimation: In such case elimination phase dependent parameters will not be reliably characterized. Hence, elimination phase dependent parameter (AUC<sub>0-inf</sub>) will be excluded from statistical analysis.
- Handling of Subjects with Non-Zero Pre-dose Concentrations:

If non-zero pre-dose concentrations occur, the following procedure will be used:

If the pre-dose concentration is less than or equal to 5% of the corresponding  $C_{max}$  value for that subject, the subject's data will be included in all PK measurements and calculations without any adjustment. If the pre-dose value is greater than 5% of the corresponding  $C_{max}$  value for that subject, the subject's data for the period in question will be excluded from the statistical evaluations (descriptive statistics for that period and ANOVA).

The following pharmacokinetic parameters for ENZ215 and EU- and US-sourced Prolia® will be computed using non-compartmental model using linear trapezoidal method:

Primary Pharmacokinetic Parameters:

C<sub>max</sub>: Maximum observed drug concentration

Area under the drug concentration-time curve from time day 0 to day 270, as

AUC<sub>0-t</sub> : calculated by linear up/log down trapezoidal summation

AUC<sub>0-inf</sub> : Area under the drug concentration-time curve from time 0 to time infinity.

Secondary Pharmacokinetic Parameters:

Partial area under the drug concentration-time curve from time 0 (Pre-dose) to

AUC<sub>0- Day 28</sub> : day 28 as calculated by linear up/log down trapezoidal summation.

Time to reach  $C_{max}$ . If the maximum value occurs at more than one time point,

 $T_{max}$ :  $t_{max}$  is defined as the first time point with this value.

 $T_{1/2}$ : The terminal elimination half-life as calculated by  $0.693/\lambda_z$ .

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




Apparent systemic clearance will be calculated using the formula:

CL/F : [Dose/AUC<sub>0-inf</sub>]

#### Analysis of Primary Pharmacokinetic Endpoints:

To demonstrate bioequivalence between ENZ215 and EU - and US-sourced Prolia® of the In-transformed pharmacokinetic parameters  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-inf}$ , Analysis of Variance (ANOVA) will be performed on the natural log (In)-transformed PK parameters ( $AUC_{0-inf}$ ,  $AUC_{0-t}$ ,  $C_{max}$ ) using Type III sum of squares, with the fixed effect of treatment using General Linear Model (PROC GLM) of SAS software. Each analysis of variance will include calculation of least square mean (LSM). Two one-sided tests procedure at 5% level of significance will be used to compare the geometric LSM values of PK parameters determined after administration of test (Treatment A) and reference products (Treatment B i.e., US Source Prolia & Treatment C i.e., EU Source Prolia).

Bioequivalence testing hypothesis as follows:

H0: 90% confidence interval (CI): lower limit < 80.00% or upper limit > 125.00% (ie, both treatments are bio-inequivalent).

H1: 90% CI: lower limit  $\geq$  80.00% and upper limit  $\leq$  125.00% (i.e., both treatments are bioequivalent).

Point estimates of the ratio of geometric least squares means of ENZ215(test)/EU sourced Prolia (Reference B), ENZ215(test)/ US sourced Prolia (Reference A), EU sourced Prolia /US sourced Prolia treatments will be calculated and reported for ln-transformed PK parameters  $C_{max}$  AUC $_{0-t}$  and AU $_{C0-\infty}$ . The inter subject variability will be calculated and reported for ln-transformed pharmacokinetic parameters  $C_{max}$  AUC $_{0-t}$  and AU $_{C0-\infty}$ .

The following treatment comparisons will be made to assess the bioequivalence between the test and each of the 2 reference treatments.

ENZ215 versus EU sourced Prolia

ENZ215 versus US sourced Prolia

The 90% CI of the geometric least squares mean ratios (ENZ215(test)/EU sourced Prolia and ENZ215/US sourced Prolia) for log-transformed primary PK parameters (AUC<sub>0-∞</sub>, AUC<sub>0-t</sub>, and C<sub>max</sub>) will be determined exponentiation of the CIs obtained for the difference between treatment least-squares means (LSM) resulting from the analyses on the ln-transformed primary PK parameters for ENZ215 versus EU

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS TP BS016 Revision 7 Reference: CS WI BS005





sourced Prolia and ENZ215 versus EU sourced Prolia.

**IIQVIA** 

The respective treatment product (ENZ215) will be concluded bioequivalent to the reference product (EU sourced Prolia and US sourced Prolia), if the 90% CI for geometric LSM ratios of ln-transformed parameters  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$  and falls within the acceptance range of 80.00% to 125.00%.

Analysis of Secondary Pharmacokinetic Endpoints:

The time to maximum observed serum concentration ( $t_{max}$ ), partial Area under curve from time 0 to 28 days (pAUC<sub>0-28days</sub>), apparent terminal half-life ( $t_{1/2}$ ), terminal rate constant ( $\lambda_z$ ), and systemic clearance (CL) as a secondary parameter will be summarized as described below.

The above PK parameters will be summarized by-treatment using n, mean, SD, %CV, minimum, median, maximum, geometric mean, and geometric %CV except that t<sub>max</sub> will be reported with n, minimum, median, and maximum only.

The In-transformed pharmacokinetic parameter of partial Area under curve from time 0 to 28 days (pAUC<sub>0-28days</sub>) will be compared between ENZ215 and Prolia using PROC TTEST of SAS software.

The non-parametric analysis (Wilcoxon-rank sum test) will be used for the comparison of  $t_{max}$  between ENZ215 and Prolia.

All Pharmacokinetic data analysis, summaries, Figures and listings will be based on the Pharmacokinetic Analysis Set.

### 17. PHARMACODYNAMIC ANALYSIS

# 17.1. Pharmacodynamic Concentrations

Subjects with partial data will be evaluated on a case-by-case basis to determine if sufficient data are available for reliable estimation of PD parameter. A listing of PD blood sample collection times as well as derived sampling time deviations will be provided.

Serum concentrations of CTX-1 will be summarized using descriptive statistics for each treatment Concentrations that are below the lower limit of quantification (BLQ) will be treated as zero for the

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


computation of descriptive statistics.

Figures of arithmetic mean concentration-time data (±SD, as appropriate) will be presented for each treatment on linear and semi-logarithmic scales. Individual subject concentration-time data will be graphically presented on linear and semi-logarithmic scales for each treatment.

Individual concentrations which are BLQ will be displayed as zero in the graphic presentations on linear scale; but will not be plotted on semi-logarithmic scale. Mean values BLQ will be displayed as 0 in the graphic presentations on linear scale but will not be plotted on semi-logarithmic scale.

### 17.2. Pharmacodynamic Parameters

For PD parameter calculations, predose samples that are BLQ will be assigned a numerical value of zero. The BLQ value may be observed during the reduction of the profile then it will be set to zero. Following BLQ values embedded between 2 quantifiable data points will be set to missing when calculating PD parameters.. Actual elapsed time from dosing will be used if a sample is collected outside the timewindow period otherwise scheduled time will be used for the final serum PD parameter calculations.

The following pharmacodynamic parameter for ENZ215 and EU- and US-sourced Prolia<sup>®</sup> will be computed using non-compartmental model using linear trapezoidal method:

Pharmacodynamic exclusion criteria:

- Criteria for exclusion of pharmacodynamics parameter of a particular subject will be as below:
  - Three consecutive missing(m) samples in the late phase may significantly influence AUEC, such subjects will not be considered for the AUEC comparison.
  - Subjects having any major protocol deviations or other clinical observations that can impact the PD.

Pharmacodynamic Parameters:

Area under the effect curve (AUEC) from time 0 to day 270 for serum CTX-1 percent

AUEC : inhibition

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


Pharmacodynamic effect for serum CTX-1 will be assessed as % reduction from baseline.

Note: % reduction from baseline serum of CTX-1 will be calculated using following formula: % reduction from baseline serum CTX-1 =[(CTX-1 (0) – CTX-1 (Ti))/CTX-1 (0)]\*100 Where CTX-1 (Ti) is the measured CTX-1 at the time Ti and CTX-1 (0) is the measured CTX-1 prior to administration of Denosumab. Here Ti (i=24, 48, 72, ...., 6456 hrs.) denotes the post dose time points at which sample has been taken. If the predose concentration is zero, then the % change cannot be calculated, and it will be considered as missing for the statistical analysis.

#### Analysis of Secondary Pharmacodynamic Endpoints:

The AUEC will be calculated as the area under the effect curve from baseline until CTX-1 values return to baseline for the first time.

An ANCOVA will be performed on the log-transformed AUEC, including treatment as a fixed effect and baseline CTX-1 value as covariate. The assessment of serum CTX-1 similarity as a secondary endpoint will be based upon the 95% confidence intervals for the ratio of the geometric means (ENZ215 and Prolia) for AUEC of baseline-corrected serum CTX-1 (i.e. % change from baseline), which have to be contained entirely within the pre-specified limits of 0.80-1.25.

All Pharmacodynamic data analysis, summaries, figures and listings will be based on the Pharmacodynamic Analysis Set.

#### 18. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the Safety Analysis Set.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified with the relevant section.

#### 18.1. Adverse Events

Adverse Events (AEs) will be coded using MedDRA, the latest version.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


after the administration of study medication. Pretreatment AEs are defined as AEs occurring prior to dosing. These events will be presented in the listing only and are not included in the tabular summary of TEAEs.

Multiple occurrences of the same TEAE in one subject during the study will be counted as multiple events in the frequency counts for adverse events. If a subject experiences more than one occurrence of the same TEAE during the trial, the subject will only be counted once using the worst severity.

See Appendix 2 for handling of partial dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, the AE will be classified by the worst case, i.e. treatment emergent.

#### **18.1.1.** All TEAEs

Incidence of TEAEs will be presented by System Organ Class (SOC) and Preferred Term (PT) and broken down further by maximum severity and relationship to study medication.

#### 18.1.1.1. SEVERITY

Severity is classed as mild/ moderate/ severe/ life threatening/ death. TEAEs starting after the first dose of study medication with a missing severity will be classified as severe. If a subject reports a TEAE more than once within that SOC/ PT, the AE with the worst-case severity will be used in the corresponding severity summaries.

#### 18.1.1.2. RELATIONSHIP TO STUDY MEDICATION

Relationship, as indicated by the Investigator, is classed as "unrelated" and "related". TEAEs with a missing relationship to study medication will be regarded as "related" to study medication. If a subject reports the same AE more than once within that SOC/ PT, the AE with the worst-case relationship to study medication will be used in the corresponding relationship summaries.

All AE tabulations will be performed by treatment. Incidence of TEAEs will be tabulated by the following:

- An overall summary across all SOC and PT, any TEAE, any related TEAE, severe, serious, leading to study discontinuation, leading to death, and TEAEs by maximum severity
- By SOC and PT

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


- By SOC and PT for related TEAEs
- By SOC, PT and Severity
- By SOC, PT and Outcome
- By SOC, PT and Seriousness (Serious = Yes or No)
- By SOC, PT and Severity for related TEAEs

### 18.1.2. TEAEs Leading to Discontinuation of Study Medication

TEAEs leading to permanent discontinuation of study medication will be identified by using the field "Action taken with study treatment = Drug withdrawal" on the AE page of the (e)CRF, and listed.

#### 18.1.3. Serious Adverse Events

Serious adverse events (SAEs) are those events recorded as "Serious" on the Adverse Events page of the (e)CRF and will be listed and summarized

### 18.1.4. Injection Site Reaction Assessment

Injection site reaction assessment will be listed including intensity grade.

### 18.2. Deaths

If any subjects die during the study as recorded on the AE page of the eCRF, the information will be presented in a data listing.

# 18.3. Laboratory Evaluations

Results from the central laboratory will be included in the reporting of this study for Hematology, Serum Chemistry and Urinalysis. A list of laboratory assessments to be included in the outputs is included in the protocol, Section 11.2.

Presentations will use units as per Celerion lab units with the conversion factor provided in Appendix 3. Quantitative laboratory measurements reported as "< X", i.e., below the lower limit of quantification (BLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for the

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

The following summaries will be provided for laboratory data:

- Actual and change from baseline by visit (for quantitative measurements)
- Listing of laboratory results outside the normal range

### 18.3.1. Laboratory Reference Ranges

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

#### 18.4. ECG Evaluations

The following ECG parameters will be reported for this study: PR, QRS, QTcB, QTcF, RR and heart rate.

- Overall assessment of ECG (Investigator's judgment):
  - o Normal
  - o Abnormal, Not Clinically Significant (ANCS)
  - o Abnormal, Clinically Significant (ACS)

The following summaries will be provided for ECG data:

- Actual and change from baseline by visit (for quantitative measurements)
- Incidence of clinically noteworthy criteria
- Listing of subjects meeting clinically noteworthy criteria

#### 18.4.1. Clinically Noteworthy ECG Criteria

Clinically noteworthy quantitative ECG measurements will be identified in accordance with the following predefined criteria:

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


- Absolute values for QTcF will be classified as:
  - $\circ$  > 450 msec and <=480 msec
  - $\circ$  > 480 msec and <=500 msec
  - $\circ$  > 500 msec
- Change from Baseline for QTcF will be classified as:
  - o Increase from baseline >30 msec and <=60 msec
  - o Increase from baseline >60 msec

### 18.5. Vital Signs

The following Vital Signs measurements will be reported for this study:

- Supine Systolic Blood Pressure (mmHg)
- Supine Diastolic Blood Pressure (mmHg)
- Supine Pulse Rate (bpm)
- Respiratory Rate (breaths/min)
- Body temperature (° C)

The following summaries will be provided for vital signs data:

• Actual and change from baseline by visit

## 18.6. Physical Examination

Physical examination results will be listed including specification of any abnormalities observed.

#### 18.7. Oral Examination

Oral examination results will be listed including specification of any abnormalities observed.

#### 18.8. COVID-19 Assessment

Results from COVID-19 testing and assessment of COVID-19 signs and symptoms will be listed.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


### 18.9. Immunogenecity Assessment

All immunogenicity data summaries will be based on the safety analysis population. Immunogenicity (ADA) including NAb data will be presented for all subjects' samples collected in data listing.

The frequency and percentage of positive ADA or NAb result will be provided. The proportion of positive ADA or NAb in each treatment group will be compared using chi-square or Fisher's exact tests. The p-value, relative risk and corresponding 95% CI will be presented.

### 19. DATA NOT SUMMARIZED OR PRESENTED

Comments will not be summarized or presented but will be available in clinical study database.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005


# 20. REFERENCES

There are no references.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005




APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

### THE LEVEL TO THE CONTROL OF THE CONT

### **IQVIA Output Conventions**

Outputs will be presented according to the IQVIA Global Biostatistics Standard Output Conventions, which is available upon request.

#### **Dates & Times**

Depending on data availability, if not otherwise specified, dates will take the format DDMMMYYYY; times will take the format hh:mm; combined dates and time will take the format DMMMYYYY/hh:mm.

## **Spelling Format**

English US.

## **Presentation of Treatment Groups**

For outputs, treatment groups will be represented as follows, as appropriate: ENZ215, US-Prolia, EU-Prolia, All Subjects (where applicable).

#### **Presentation of Visits**

For outputs, visits will be represented as collected on eCRF, as appropriate.

## Listings

All listings will be ordered by the following (unless otherwise indicated in the template):

- Treatment
- Subject number
- Date and Time (where applicable)
- For listings where non-randomized subjects are included (e.g. screen failures, if applicable), these will appear in a category after the randomized treatment groups labeled 'Not Randomized'

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




# APPENDIX 2. PARTIAL DATE CONVENTIONS

Imputed dates will NOT be presented in the listings.

# **Algorithm for Treatment Emergence of Adverse Events:**

| START DATE/TIME | STOP<br>DATE/TIME | ACTION |
|---|---|---|
| Known | Known/Partial/<br>Missing | If start date/time < study med start date/time, then not TEAE If start date/time >= study med start date/time, then TEAE |
| Partial, but known components show that it cannot be on or after study med start date | Known/Partial/<br>Missing | Not TEAE |
| Partial, could be on or after study med start date OR Missing | Known | If stop date/time < study med start date/time, then not TEAE If stop date/time >= study med start date/time, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date/time < study med start date/time, then not TEAE If stop date/time >= study med start date/time, then TEAE |
| | Missing | Assumed TEAE |

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-Document:

DEN1\_HAB89093\Biostatistics\Documentation\SAP

1.0 Author: Ashutosh Ranjan, Piyushkumar Jogani Version Number:


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS WI BS005



# **Algorithm for Prior / Concomitant Medications:**

| START<br>DATE/TIME | STOP<br>DATE/TIME | ACTION |
|---|---|---|
| Known | Known | If stop date/time < study med start date/time, assign as prior If stop date/time >= study med start date/time, assign as concomitant |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date/time < study med start date/time, assign as prior If stop date/time >= study med start date/time, assign as concomitant |
| | Missing | If stop date is missing could never be assumed a prior medication assign as concomitant |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date/time < study med start date/time, assign as prior If stop date/time >= study med start date/time, assign as concomitant |
| | Partial | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown) and impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date/time < study med start date/time, assign as prior If stop date/time >= study med start date/time, assign as concomitant |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




| START | STOP | ACTION |
|---|---|---|
| DATE/TIME | DATE/TIME | |
| | Missing | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date is missing could never be assumed a prior medication, assign as concomitant |
| Missing | Known | If stop date/time < study med start date/time, assign as prior If stop date/time >= study med start date/time, assign as concomitant |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date/time < study med start date/time, assign as prior If stop date/time >= study med start date/time, assign as concomitant |
| | Missing | Assign as concomitant |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

**IIQVIA** 





| | MTZ | COMAC | Celerion | Conversion factor | Conversion units |
|---|---|---|---|---|---|
| Lab tests | Units | Units | Units | | |
| Alanine<br>Aminotransferase | U/L | U/L | U/L | | |
| Albumin | g/dL | g/L | g/L | 10.0 | Conventional unit to SI unit |
| Alkaline phosphatase | U/L | U/L | U/L | | |
| Aspartate<br>Aminotransferase | U/L | U/L | U/L | | |
| Bilirubin, total | mg/dL | umol/L | umol/L | 17.1 | Conventional unit to SI unit |
| Chloride | mmol/L | mmol/L | mmol/L | | |
| Creatinine | mg/dL | umol/L | umol/L | 88.4 | Conventional unit to SI unit |
| Magnesium | mg/dL | mmol/L | mmol/L | 0.411 | Conventional unit to SI unit |
| Phosphate<br>(Phosphorus) | mg/dL | mmol/L | mmol/L | 0.323 | Conventional unit to SI unit |
| Potassium | mmol/L | mmol/L | mmol/L | | |
| Protein, Total | g/dL | g/L | g/L | 10.0 | Conventional unit to SI unit |
| Sodium | mmol/L | mmol/L | mmol/L | | |
| Blood Urea Nitrogen | mg/dL | mmol/L | mmol/L | 0.357 | Conventional unit to SI unit |
| | mmol/L | | | | |
| Glucose | mg/dL | mmol/L | mmol/L | 0.0555 | Conventional unit to SI unit |
| | mmol/L | | | | |
| Calcium | mg/dL | mmol/L | mmol/L | 0.25 | Conventional unit to SI unit |
| Albumin adjusted calcium | mg/dL | mmol/L | mmol/L | 1 mg/dl= 0.2495<br>mmol/L | Conventional unit<br>to SI unit |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

 $Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 \ IQVIA. \ All \ rights \ reserved. \ The \ contents \ of this \ document \ are \ confidential \ and \ proprietary \ to \ IQVIA \ Holdings \ Inc. \ and \ its \ subsidiaries. \ Unauthorized \ use, \ disclosure \ or \ reproduction \ is \ strictly \ prohibited.$ 




| | MTZ | COMAC | Celerion | Conversion factor | Conversion units |
|---|---|---|---|---|---|
| Lab tests | Units | Units | Units | | |
| Red Blood Cell Count<br>(Total) | 10**12/L | T/L | X 10 <sup>12</sup> /L | | |
| Hemoglobin | g/dL | | g/dL | 10.0 | SI unit to<br>Conventional unit |
| White Blood Cell Count (Total) | 10**9/L | G/L | X 10 <sup>9</sup> /L | | |
| Platelets | 10**9/L | G/L | X 10 <sup>9</sup> /L | | |
| Neutrophils, Absolute<br>Count | 10**9/L | G/L | X 10 <sup>9</sup> /L | | |
| Lymphocytes,<br>Absolute Count | 10**9/L | | X 10 <sup>9</sup> /L | | |
| Monocytes, Absolute<br>Count | 10**9/L | | X 10 <sup>9</sup> /L | | |
| Eosinophils, Absolute<br>Count | 10**9/L | | X 10 <sup>9</sup> /L | | |
| Basophils, Absolute<br>Count | 10**9/L | G/L | X 10 <sup>9</sup> /L | | |
| Neutrophils (Rel, %) | % | % | % | | |
| Lymphocytes (Rel, %) | % | % | % | | |
| Monocytes (Rel, %) | % | % | % | | |
| Eosinophils (Rel, %) | % | % | % | | |
| Basophils (Rel, %) | % | % | % | | |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\Alkem\Denosumab\ALK22ENZ215-

DEN1\_HAB89093\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

# **DocuSign**

#### **Certificate Of Completion**

Envelope Id: 6B27F3E532A5491D929BB13B6DEBDFB0

Subject: Complete with Docusign: Alkem\_ALK22ENZ215\_DEN1\_SAP\_v1.0\_Alkem\_21Jun2024.docx

Project Code (Enter 0 for non-billable projects): HAB89093

IQVIA ID (Login ID): 802036

**Business Unit:** 

DSSR

Source Envelope:

Document Pages: 41Signatures: 5Envelope Originator:Certificate Pages: 5Initials: 0Ashutosh RanjanAutoNav: EnabledOne IMS Way

Envelopeld Stamping: Disabled

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Plymouth Meeting, 19462 Ashutosh.Ranjan@quintiles.com

IP Address: 162.44.245.32

Sent: 21-Jun-2024 | 21:12

Viewed: 24-Jun-2024 | 14:35

Signed: 24-Jun-2024 | 14:36

### **Record Tracking**

Status: Original

21-Jun-2024 | 21:09

Holder: Ashutosh Ranjan

Ashutosh.Ranjan@quintiles.com

Location: DocuSign

**Timestamp** 

Status: Completed

#### **Signer Events**

Ashutosh Ranjan

ashutosh.ranjan@quintiles.com

Statistical Scientist

QVIA

Security Level: Email, Account Authentication

(Required)

Signature

Ashvtosh Panjan

Signature Adoption: Pre-selected Style

Signature ID:

55DBAAC8-8C76-431C-8552-29B736B6AF8D

Using IP Address: 162.44.245.32

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I am the author of this document
I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Piyushkumar Jogani

Piyushkumar.Jogani@premier-research.com

Biostatistician

Premier Research

Security Level: Email, Account Authentication

(Required)

Piyushkumar Jogani

Signature Adoption: Pre-selected Style

Signature ID:

D1E3500D-6D85-4D03-80A0-B51EE2459E48

Using IP Address: 49.36.69.78

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 24-Jun-2024 | 04:25

ID: 3784639d-dd67-4222-9b8f-c395d0c1201b

Sent: 21-Jun-2024 | 21:12 Viewed: 24-Jun-2024 | 04:25 Signed: 24-Jun-2024 | 10:23 Signer Events

Vinayaka Shahavi vinayaka.shahavi@alkem.com General Manager-Clinical Research Security Level: Email, Account Authentication

(Required)

**Signature** 

DocuSigned by Vinayaka Shahavi



I approve this document June 22, 2024 | 12:03:55 AM PDT **Timestamp** 

Sent: 21-Jun-2024 | 21:12

Viewed: 22-Jun-2024 | 08:01

Signed: 22-Jun-2024 | 08:05

\_\_\_\_\_D3E46A69468042D8B98B6A970A59FD0A

Signature Adoption: Pre-selected Style

Signature ID:

D3E46A69-4680-42D8-B98B-6A970A59FD0A

Using IP Address: 1.38.220.10

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 22-Jun-2024 | 08:01

ID: 053df98d-5419-4a95-b485-0346dc87c87a

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 21-Jun-2024 21:12<br>22-Jun-2024 08:01<br>22-Jun-2024 08:05<br>24-Jun-2024 14:36 |
| Payment Events | Status | Timestamps |

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents will be sent to you electronically**

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### **How to contact IOVIA:**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

## 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

### 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

### 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.